CLINICAL TRIAL: NCT03106636
Title: Randomized Trial of KEEP-P, a Preventive Intervention for Foster Preschoolers
Brief Title: Trial of KEEP-P, a Preventive Intervention for Foster Preschoolers (KEEP-P)
Acronym: KEEP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Phil Fisher, Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06112013.016
Record Dates: First submitted 2015-06-04; First posted 2017-04-10 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Child Behavior
Keywords: Preschool-aged; Foster children; child welfare; Fostercare; Parent training; early adversity; curriculum based; early intervention; preschool; foster placement disruptions; manualized intervention; group based intervention; high-risk children
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KEEP-P (Active Comparator): Caregivers are randomly assigned to one of two groups. The KEEP-P group completes a basic version of the curriculum. The intervention content is delivered by a KEEP-P group facilitator in a 2-hour weekly group format. Duration of the program is 12 weeks.
  Interventions: Behavioral: KEEP-P
- KEEP-P+ (Experimental): Caregivers are randomly assigned to one of two groups. The KEEP-P+ group completes an augmented version of the intervention with curriculum that includes the addition of information about recent findings in early brain development and a video coaching component based on the Filming Interactions to Nurture Development (FIND) program. The intervention content is delivered by a KEEP-P group facilitator in a 2-hour weekly group format. Duration of the program is 12 weeks.
  Interventions: Behavioral: KEEP-P+

INTERVENTIONS:
Behavioral: KEEP-P — The KEEP-P program is a low-cost, manualized, group-based intervention for caregivers of preschool aged children. This trial is evaluating 2 versions of the intervention. KEEP-P is a basic version that employs a curriculum of 12 weekly psychoeducational caregiver support groups Across four waves of data collection (baseline, post-intervention, and 12 and 18 months post-baseline), we will examine the extent to which this intervention condition shows improved parenting, reduced rates of disrupted placements, and improved child outcomes.
  Arms: KEEP-P
Behavioral: KEEP-P+ — The KEEP-P program is a low-cost, manualized, group-based intervention for caregivers of preschool aged children. This trial is evaluating 2 versions of the intervention. KEEP-P+ is an augmented version that consists of the caregiver support groups with extended curriculum including information about recent findings in early brain development and the elements of the Filming Interactions to Nurture Development video coaching program. Across four waves of data collection (baseline, post-intervention, and 12 and 18 months post-baseline), we will examine the extent to which this intervention condition show improved parenting, reduced rates of disrupted placements, and improved child outcomes.
  Arms: KEEP-P+

SUMMARY:
Randomized Trial of KEEP-P, a Preventive Intervention for Foster Preschoolers (KEEP-P). The goal of the proposed study is to conduct a randomized clinical trial of a new, low-cost, manualized, group-based intervention for preschoolers and their caregivers. The investigators will examine the extent to which the two intervention conditions show improved parenting, reduced rates of disrupted placements, and improved child outcomes.

DETAILED DESCRIPTION:
Randomized Trial of KEEP-P, a Preventive Intervention for Foster Preschoolers (KEEP-P).

Preschool-aged foster and other high-risk children are at increased risk for numerous negative outcomes. However, there is very limited use of evidence-based interventions for these young children. Major barriers to progress in this area include a lack of available evidence-based programs for high-risk children across the preschool years and the tendency for the few existing evidence-based interventions to be resource intensive in terms of funding and the level of staff expertise required to be implemented with fidelity. Readily scalable, evidence-based interventions for foster and other high-risk preschoolers are clearly needed to reduce the widespread disparities. The goal of the proposed study is to conduct a randomized clinical trial of a new, low-cost, manualized, group-based intervention for caregivers of preschool aged children. The investigators propose to evaluate two versions of the intervention: (a) a basic version that employs a curriculum consisting of 12 weekly psychoeducational caregiver support groups and (b) an augmented version that consists of the caregiver support groups with extended curriculum including with the addition of information about recent findings in early brain development and the elements of the Filming Interactions to Nurture Development (FIND) video coaching program. Across four waves of data collection (baseline, immediately postintervention, and 12 and 18 months postbaseline), the investigators will examine the extent to which the two intervention conditions show improved parenting, reduced rates of disrupted placements, and improved child outcomes. The investigators will conduct multivariate modeling to examine mediating mechanisms underlying the hypothesized immediate and longer- term intervention effects.

Finally, the investigators will conduct a comprehensive economic evaluation to examine the incremental costs associated with implementing the intervention and the benefits realized in the intervention conditions in terms of increased positive outcomes for children.

ELIGIBILITY:
Inclusion Criteria:

* Preschool-aged foster children
* Preschool-aged children referred to early intervention/childhood special education services

Exclusion Criteria:

* Children will be excluded from recruitment if they or their primary caregiver are not sufficiently fluent in English to complete the assessment or if it is determined that the child would not be able to complete the assessment procedures due to a severe developmental, medical, or physical disorder.

Ages: 30 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 442 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Fisher, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD data will be shared with other researchers upon completion of the data set as well as completion of a data sharing agreement.

REFERENCES:
- [Background] Aarons GA, Brown SA, Hough RL, Garland AF, Wood PA. Prevalence of adolescent substance use disorders across five sectors of care. J Am Acad Child Adolesc Psychiatry. 2001 Apr;40(4):419-26. doi: 10.1097/00004583-200104000-00010. PMID 11314567
- [Background] Barth, R. P., Scarborough, A. A., Lloyd, C. E., Losby, J. L., Casanueva, C., & Mann, T. (2007). Developmental status and early intervention service needs of maltreated children. Washington, DC: U.S. Department of Health and Human Services, Office of the Assistant Secretary for Planning and Evaluation.
- [Background] Bonomi AE, Cannon EA, Anderson ML, Rivara FP, Thompson RS. Association between self-reported health and physical and/or sexual abuse experienced before age 18. Child Abuse Negl. 2008 Jul;32(7):693-701. doi: 10.1016/j.chiabu.2007.10.004. Epub 2008 Jul 7. PMID 18602692
- [Background] Chartier MJ, Walker JR, Naimark B. Separate and cumulative effects of adverse childhood experiences in predicting adult health and health care utilization. Child Abuse Negl. 2010 Jun;34(6):454-64. doi: 10.1016/j.chiabu.2009.09.020. Epub 2010 Apr 20. PMID 20409586
- [Background] English DJ, Graham JC, Litrownik AJ, Everson M, Bangdiwala SI. Defining maltreatment chronicity: are there differences in child outcomes? Child Abuse Negl. 2005 May;29(5):575-95. doi: 10.1016/j.chiabu.2004.08.009. PMID 15970326
- [Background] Fantuzzo, J. W., & Perlman, S. M. (2007). The unique impact of out-of-home placement and the mediating effects of child maltreatment and homelessness on early school success. Children and Youth Services Review, 29, 941-960.
- [Background] Fisher, P. A., & Gunnar, M. R. (2010). Early life stress as a risk factor for disease in childhood. In R. A. Lanius, E. Vermetten & C. Pain (Eds.), The impact of early life trauma on health and disease (pp. 133-141). Cambridge, UK: Cambridge University Press.
- [Background] Garland AF, Hough RL, McCabe KM, Yeh M, Wood PA, Aarons GA. Prevalence of psychiatric disorders in youths across five sectors of care. J Am Acad Child Adolesc Psychiatry. 2001 Apr;40(4):409-18. doi: 10.1097/00004583-200104000-00009. PMID 11314566
- [Background] Kaplow JB, Widom CS. Age of onset of child maltreatment predicts long-term mental health outcomes. J Abnorm Psychol. 2007 Feb;116(1):176-87. doi: 10.1037/0021-843X.116.1.176. PMID 17324028
- [Background] Keiley MK, Howe TR, Dodge KA, Bates JE, Petti GS. The timing of child physical maltreatment: a cross-domain growth analysis of impact on adolescent externalizing and internalizing problems. Dev Psychopathol. 2001 Fall;13(4):891-912. PMID 11771913
- [Background] Lewis DO, Pincus JH, Lovely R, Spitzer E, Moy E. Biopsychosocial characteristics of matched samples of delinquents and nondelinquents. J Am Acad Child Adolesc Psychiatry. 1987 Sep;26(5):744-52. doi: 10.1097/00004583-198709000-00022. No abstract available. PMID 3667506
- [Background] McCluskey, C. P., Krohn, M. D., Lizotte, A. J., & Rodriguez, M. L. (2002). Early substance use and school achievement: An examination of Latino, White, and African American youth. Journal of Drug Issues, 32, 921-943.
- [Background] Pawlby SJ, Mills A, Quinton D. Vulnerable adolescent girls: opposite-sex relationships. J Child Psychol Psychiatry. 1997 Nov;38(8):909-20. doi: 10.1111/j.1469-7610.1997.tb01610.x. PMID 9413791
- [Background] Schneiderman JU, Leslie LK, Arnold-Clark JS, McDaniel D, Xie B. Pediatric health assessments of young children in child welfare by placement type. Child Abuse Negl. 2011 Jan;35(1):29-39. doi: 10.1016/j.chiabu.2010.06.007. PMID 21316106
- [Background] Tarren-Sweeney M, Hazell P. Mental health of children in foster and kinship care in New South Wales, Australia. J Paediatr Child Health. 2006 Mar;42(3):89-97. doi: 10.1111/j.1440-1754.2006.00804.x. PMID 16509906
- [Background] Anderson LM, Shinn C, Fullilove MT, Scrimshaw SC, Fielding JE, Normand J, Carande-Kulis VG; Task Force on Community Preventive Services. The effectiveness of early childhood development programs. A systematic review. Am J Prev Med. 2003 Apr;24(3 Suppl):32-46. doi: 10.1016/s0749-3797(02)00655-4. PMID 12668197
- [Background] Ramey CT, Ramey SL. Early intervention and early experience. Am Psychol. 1998 Feb;53(2):109-20. doi: 10.1037//0003-066x.53.2.109. PMID 9491742
- [Background] Aos, S., Lieb, R., Mayfield, J., Miller, M., & Pennucci, A. (2004). Benefits and costs of prevention and early intervention programs for youth. Olympia, WA: Washington State Institute for Public Policy.
- [Background] Heckman JJ. Skill formation and the economics of investing in disadvantaged children. Science. 2006 Jun 30;312(5782):1900-2. doi: 10.1126/science.1128898. PMID 16809525
- [Background] Price, J. M., Chamberlain, P., Landsverk, J., & Reid, J. (2009). KEEP foster-parent training intervention: Model description and effectiveness. Child and Family Social Work, 14, 233-242.
- [Background] U.S. Department of Health and Human Services. (2011). The AFCARS Report: Preliminary FY 2010 Estimates as of June 2011. Washington, DC: Author.
- [Background] Kessler RC, Pecora PJ, Williams J, Hiripi E, O'Brien K, English D, White J, Zerbe R, Downs AC, Plotnick R, Hwang I, Sampson NA. Effects of enhanced foster care on the long-term physical and mental health of foster care alumni. Arch Gen Psychiatry. 2008 Jun;65(6):625-33. doi: 10.1001/archpsyc.65.6.625. PMID 18519820
- [Background] Cullen, J. P., Ownbey, J. B., & Ownbey, M. A. (2010). The effects of the Healthy Families America home visitation program on parenting attitudes and practices and child social and emotional competence. Child and Adolescent Social Work Journal, 27, 335-354.
- [Background] Eckenrode J, Campa M, Luckey DW, Henderson CR Jr, Cole R, Kitzman H, Anson E, Sidora-Arcoleo K, Powers J, Olds D. Long-term effects of prenatal and infancy nurse home visitation on the life course of youths: 19-year follow-up of a randomized trial. Arch Pediatr Adolesc Med. 2010 Jan;164(1):9-15. doi: 10.1001/archpediatrics.2009.240. PMID 20048236
- [Background] Howard KS, Brooks-Gunn J. The role of home-visiting programs in preventing child abuse and neglect. Future Child. 2009 Fall;19(2):119-46. doi: 10.1353/foc.0.0032. PMID 19719025
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Dubowitz, H. (1990). The physical and mental health and educational status of children placed with relatives: Final report. Baltimore, MD: Department of Pediatrics, School of Medicine.
- [Background] Pears K, Fisher PA. Developmental, cognitive, and neuropsychological functioning in preschool-aged foster children: associations with prior maltreatment and placement history. J Dev Behav Pediatr. 2005 Apr;26(2):112-22. doi: 10.1097/00004703-200504000-00006. PMID 15827462
- [Background] Simms MD. The foster care clinic: a community program to identify treatment needs of children in foster care. J Dev Behav Pediatr. 1989 Jun;10(3):121-8. PMID 2473095
- [Background] Leslie LK, Gordon JN, Meneken L, Premji K, Michelmore KL, Ganger W. The physical, developmental, and mental health needs of young children in child welfare by initial placement type. J Dev Behav Pediatr. 2005 Jun;26(3):177-85. doi: 10.1097/00004703-200506000-00003. PMID 15956866
- [Background] Brooks, D., & Barth, R. P. (1998). Characteristics and outcomes of drug-exposed and non drug-exposed children in kinship and non-relative foster care. Children and Youth Services Review, 20, 475-501.
- [Background] Colton, M., Heath, A., & Aldgate, J. (1995). Factors which influence the educational attainment of children in foster family care. Community Alternatives: International Journal of Family Care, 7, 15-36.
- [Background] Dumaret A. IQ, scholastic performance and behaviour of sibs raised in contrasting environments. J Child Psychol Psychiatry. 1985 Jul;26(4):553-80. doi: 10.1111/j.1469-7610.1985.tb01641.x. PMID 4019617
- [Background] Pears KC, Fisher PA, Bruce J, Kim HK, Yoerger K. Early elementary school adjustment of maltreated children in foster care: the roles of inhibitory control and caregiver involvement. Child Dev. 2010 Sep-Oct;81(5):1550-64. doi: 10.1111/j.1467-8624.2010.01491.x. PMID 20840240
- [Background] Stein, E. (1997). Teachers' assessments of children in foster care. Developmental Disabilities Bulletin, 25, 1-17.
- [Background] Zima, B. T., Bussing, R., Freeman, S., Yang, X., Belin, T. R., & Forness, S. R. (2000). Behavior problems, academic skill delays and school failure among school-aged children in foster care: Their relationship to placement characteristics. Journal of Child and Family Studies, 9, 87-103.
- [Background] Goerge, R. M., Van Voorhis, J., Grant, S., Casey, K., & Robinson, M. (1992). Special-education experiences of foster children: An empirical study. Child Welfare: Journal of Policy, Practice, and Program, 71, 419-437.
- [Background] Sawyer RJ, Dubowitz H. School performance of children in kinship care. Child Abuse Negl. 1994 Jul;18(7):587-97. doi: 10.1016/0145-2134(94)90085-x. PMID 7522940
- [Background] Smith, D. K., Stormshak, E., Chamberlain, P., & Whaley, R. B. (2001). Placement disruption in treatment foster care. Journal of Emotional and Behavioral Disorders, 9, 200-205.
- [Background] Berger, L. M., Bruch, S. K., Johnson, E. I., James, S., & Rubin, D. (2009). Estimating the
- [Background] Hussey DL, Guo S. Characteristics and trajectories of treatment foster care youth. Child Welfare. 2005 Jul-Aug;84(4):485-506. PMID 16117260
- [Background] Newton RR, Litrownik AJ, Landsverk JA. Children and youth in foster care: distangling the relationship between problem behaviors and number of placements. Child Abuse Negl. 2000 Oct;24(10):1363-74. doi: 10.1016/s0145-2134(00)00189-7. PMID 11075702
- [Background] Dozier M, Bick J. Changing caregivers: coping with early adversity. Pediatr Ann. 2007 Apr;36(4):205-8. doi: 10.3928/0090-4481-20070401-09. No abstract available. PMID 17469300
- [Background] Dozier, M., & Rutter, M. (2008). Challenges to the development of attachment relationships faced by young children in foster and adoptive care. In J. Cassidy, P. R. Shaver (Eds.), Handbook of attachment: Theory, research, and clinical applications (2nd ed., pp. 698-717). New York, NY: Guilford Press.
- [Background] Zeanah CH, Shauffer C, Dozier M. Foster care for young children: why it must be developmentally informed. J Am Acad Child Adolesc Psychiatry. 2011 Dec;50(12):1199-201. doi: 10.1016/j.jaac.2011.08.001. No abstract available. PMID 22115138
- [Background] Effects of Multidimensional Treatment Foster Care for Preschoolers (MTFC-P) on Reducing Permanent Placement Failures Among Children With Placement Instability. Child Youth Serv Rev. 2009 May;31(5):541-546. doi: 10.1016/j.childyouth.2008.10.012. PMID 19430545
- [Background] Ward, H., & Holmes, L. (2008). Calculating the costs of local authority care for children with contrasting needs. Child and Family Social Work, 13, 80-90.
- [Background] Guralnick MJ. Effectiveness of early intervention for vulnerable children: a developmental perspective. Am J Ment Retard. 1998 Jan;102(4):319-45. doi: 10.1352/0895-8017(1998)1022.0.co;2. PMID 9475942
- [Background] Farmer, E. M. Z., Burns, B. J., Wagner, H. R., Murray, M., & Southerland, D. G. (2010). Enhancing
- [Background] Price JM, Chamberlain P, Landsverk J, Reid JB, Leve LD, Laurent H. Effects of a foster parent training intervention on placement changes of children in foster care. Child Maltreat. 2008 Feb;13(1):64-75. doi: 10.1177/1077559507310612. PMID 18174349
- [Background] Nilsen W. Fostering futures: a preventive intervention program for school-age children in foster care. Clin Child Psychol Psychiatry. 2007 Jan;12(1):45-63. doi: 10.1177/1359104507071055. PMID 17378079
- [Background] Fisher, P. A., Ellis, B. H., & Chamberlain, P. (1999). Early Intervention Foster Care: A model for preventing risk in young children who have been maltreated. Children's Services: Social Policy, Research, and Practice, 2, 159-182.
- [Background] Fisher PA, Gunnar MR, Chamberlain P, Reid JB. Preventive intervention for maltreated preschool children: impact on children's behavior, neuroendocrine activity, and foster parent functioning. J Am Acad Child Adolesc Psychiatry. 2000 Nov;39(11):1356-64. doi: 10.1097/00004583-200011000-00009. PMID 11068890
- [Background] Fisher PA, Burraston B, Pears K. The early intervention foster care program: permanent placement outcomes from a randomized trial. Child Maltreat. 2005 Feb;10(1):61-71. doi: 10.1177/1077559504271561. PMID 15611327
- [Background] Fisher PA, Stoolmiller M. Intervention effects on foster parent stress: associations with child cortisol levels. Dev Psychopathol. 2008 Summer;20(3):1003-21. doi: 10.1017/S0954579408000473. PMID 18606041
- [Background] Fisher PA, Gunnar MR, Dozier M, Bruce J, Pears KC. Effects of therapeutic interventions for foster children on behavioral problems, caregiver attachment, and stress regulatory neural systems. Ann N Y Acad Sci. 2006 Dec;1094:215-25. doi: 10.1196/annals.1376.023. PMID 17347353
- [Background] Fisher PA, Kim HK. Intervention effects on foster preschoolers' attachment-related behaviors from a randomized trial. Prev Sci. 2007 Jun;8(2):161-70. doi: 10.1007/s11121-007-0066-5. Epub 2007 Mar 6. PMID 17340186
- [Background] Dozier, M., Bick, J., & Bernard, K. (2011). Attachment-based treatment for young, vulnerable children. In J. D. Osofsky, A. F. Lieberman (Eds.), Clinical work with traumatized young children (pp. 75-95). New York, NY: Guilford Press.
- [Background] Dozier, M., Higley, E., Albus, K. E., & Nutter, A. (2002). Intervening with foster infants' caregivers: Targeting three critical needs. Infant Mental Health Journal, 23, 541-554.
- [Background] Dozier, M., Peloso, E., Lindhiem, O., Gordon, M. K., Manni, M., Sepulveda, S., … Levine, S. (2006). Developing evidence-based interventions for foster children: An example of a randomized clinical trial with infants and toddlers. Journal of Social Issues, 62, 767-785.
- [Background] Dozier M, Lindhiem O, Lewis E, Bick J, Bernard K, Peloso E. Effects of a Foster Parent Training Program on Young Children's Attachment Behaviors: Preliminary Evidence from a Randomized Clinical Trial. Child Adolesc Social Work J. 2009 Aug;26(4):321-332. doi: 10.1007/s10560-009-0165-1. PMID 22065891
- [Background] Dozier M, Peloso E, Lewis E, Laurenceau JP, Levine S. Effects of an attachment-based intervention on the cortisol production of infants and toddlers in foster care. Dev Psychopathol. 2008 Summer;20(3):845-59. doi: 10.1017/S0954579408000400. PMID 18606034
- [Background] Dorsey S, Farmer EM, Barth RP, Greene K, Reid J, Landsverk J. Current Status and Evidence Base of Training for Foster and Treatment Foster Parents. Child Youth Serv Rev. 2008 Dec 1;30(12):1403-1416. doi: 10.1016/j.childyouth.2008.04.008. No abstract available. PMID 21647272
- [Background] Byford, S., & Sefton, T. (2003). Economic evaluation of complex health and social care interventions. National Institute Economic Review, 186, 98-108.
- [Background] Corso PS, Fertig AR. The economic impact of child maltreatment in the United States: are the estimates credible? Child Abuse Negl. 2010 May;34(5):296-304. doi: 10.1016/j.chiabu.2009.09.014. Epub 2010 Mar 27. No abstract available. PMID 20347486
- [Background] Corso PS, Lutzker JR. The need for economic analysis in research on child maltreatment. Child Abuse Negl. 2006 Jul;30(7):727-38. doi: 10.1016/j.chiabu.2005.12.006. Epub 2006 Jul 18. No abstract available. PMID 16854463
- [Background] Sefton, T. A. J. (2003). Economic evaluation in the social welfare field. Evaluation, 9, 73-91.
- [Background] Charles JM, Bywater T, Edwards RT. Parenting interventions: a systematic review of the economic evidence. Child Care Health Dev. 2011 Jul;37(4):462-74. doi: 10.1111/j.1365-2214.2011.01217.x. Epub 2011 Mar 6. PMID 21375566
- [Background] Bywater T, Hutchings J, Linck P, Whitaker C, Daley D, Yeo ST, Edwards RT. Incredible Years parent training support for foster carers in Wales: a multi-centre feasibility study. Child Care Health Dev. 2011 Mar;37(2):233-43. doi: 10.1111/j.1365-2214.2010.01155.x. Epub 2010 Sep 21. PMID 20854449
- [Background] Lynch FL, Dickerson JF, Saldana L, Fisher PA. Incremental Net Benefit of Early Intervention for Preschool-Aged Children with Emotional and Behavioral Problems in Foster Care. Child Youth Serv Rev. 2014 Jan;36:213-219. doi: 10.1016/j.childyouth.2013.11.025. Epub 2013 Dec 5. PMID 29097828
- [Background] Lynch FL, Dickerson JF, Clarke G, Vitiello B, Porta G, Wagner KD, Emslie G, Asarnow JR Jr, Keller MB, Birmaher B, Ryan ND, Kennard B, Mayes T, DeBar L, McCracken JT, Strober M, Suddath RL, Spirito A, Onorato M, Zelazny J, Iyengar S, Brent D. Incremental cost-effectiveness of combined therapy vs medication only for youth with selective serotonin reuptake inhibitor-resistant depression: treatment of SSRI-resistant depression in adolescents trial findings. Arch Gen Psychiatry. 2011 Mar;68(3):253-62. doi: 10.1001/archgenpsychiatry.2011.9. PMID 21383263
- [Background] Lynch FL, Striegel-Moore RH, Dickerson JF, Perrin N, Debar L, Wilson GT, Kraemer HC. Cost-effectiveness of guided self-help treatment for recurrent binge eating. J Consult Clin Psychol. 2010 Jun;78(3):322-33. doi: 10.1037/a0018982. PMID 20515208
- [Background] Lynch FL, Hornbrook M, Clarke GN, Perrin N, Polen MR, O'Connor E, Dickerson J. Cost-effectiveness of an intervention to prevent depression in at-risk teens. Arch Gen Psychiatry. 2005 Nov;62(11):1241-8. doi: 10.1001/archpsyc.62.11.1241. PMID 16275811
- [Background] Gunnar MR, Fisher PA; Early Experience, Stress, and Prevention Network. Bringing basic research on early experience and stress neurobiology to bear on preventive interventions for neglected and maltreated children. Dev Psychopathol. 2006 Summer;18(3):651-77. PMID 17152395
- [Background] Eddy JM, Chamberlain P. Family management and deviant peer association as mediators of the impact of treatment condition on youth antisocial behavior. J Consult Clin Psychol. 2000 Oct;68(5):857-863. doi: 10.1037/0022-006X.68.5.857. PMID 11068971
- [Background] Leve LD, Chamberlain P, Reid JB. Intervention outcomes for girls referred from juvenile justice: effects on delinquency. J Consult Clin Psychol. 2005 Dec;73(6):1181-5. doi: 10.1037/0022-006X.73.6.1181. PMID 16392991
- [Background] Meldrum ML. A brief history of the randomized controlled trial. From oranges and lemons to the gold standard. Hematol Oncol Clin North Am. 2000 Aug;14(4):745-60, vii. doi: 10.1016/s0889-8588(05)70309-9. PMID 10949771
- [Background] Madon T, Hofman KJ, Kupfer L, Glass RI. Public health. Implementation science. Science. 2007 Dec 14;318(5857):1728-9. doi: 10.1126/science.1150009. No abstract available. PMID 18079386
- [Background] Embry DD, Biglan A. Evidence-based kernels: fundamental units of behavioral influence. Clin Child Fam Psychol Rev. 2008 Sep;11(3):75-113. doi: 10.1007/s10567-008-0036-x. PMID 18712600
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Chamberlain P, Price J, Reid J, Landsverk J. Cascading implementation of a foster and kinship parent intervention. Child Welfare. 2008;87(5):27-48. PMID 19402358
- [Background] Beers SR, De Bellis MD. Neuropsychological function in children with maltreatment-related posttraumatic stress disorder. Am J Psychiatry. 2002 Mar;159(3):483-6. doi: 10.1176/appi.ajp.159.3.483. PMID 11870018
- [Background] Blair C. Stress and the Development of Self-Regulation in Context. Child Dev Perspect. 2010 Dec;4(3):181-188. doi: 10.1111/j.1750-8606.2010.00145.x. PMID 21779305
- [Background] Blair C, Granger DA, Willoughby M, Mills-Koonce R, Cox M, Greenberg MT, Kivlighan KT, Fortunato CK; FLP Investigators. Salivary cortisol mediates effects of poverty and parenting on executive functions in early childhood. Child Dev. 2011 Nov-Dec;82(6):1970-84. doi: 10.1111/j.1467-8624.2011.01643.x. Epub 2011 Oct 25. PMID 22026915
- [Background] Blair, C., & Ursache, A. (2011). A bidirectional model of executive functions and self-regulation. In R. F. Baumeister and K. D. Vohs (Eds.), Handbook of self-regulation: Research, theory, and applications (2nd ed., pp. 300-320): New York, NY: Guilford Press.
- [Background] De Bellis MD, Thomas LA. Biologic findings of post-traumatic stress disorder and child maltreatment. Curr Psychiatry Rep. 2003 Jun;5(2):108-17. doi: 10.1007/s11920-003-0027-z. PMID 12685990
- [Background] McEwen BS. Protection and damage from acute and chronic stress: allostasis and allostatic overload and relevance to the pathophysiology of psychiatric disorders. Ann N Y Acad Sci. 2004 Dec;1032:1-7. doi: 10.1196/annals.1314.001. PMID 15677391
- [Background] Rhoades BL, Greenberg MT, Lanza ST, Blair C. Demographic and familial predictors of early executive function development: contribution of a person-centered perspective. J Exp Child Psychol. 2011 Mar;108(3):638-62. doi: 10.1016/j.jecp.2010.08.004. Epub 2010 Sep 9. PMID 20828709
- [Background] Bruce J, McDermott JM, Fisher PA, Fox NA. Using behavioral and electrophysiological measures to assess the effects of a preventive intervention: a preliminary study with preschool-aged foster children. Prev Sci. 2009 Jun;10(2):129-40. doi: 10.1007/s11121-008-0115-8. PMID 19030992
- [Background] Howse, R. B., Calkins, S. D., Anastopoulos, A. D., Keane, S. P., & Shelton, T. L. (2003). Regulatory contributors to children's kindergarten acheivement. Early Education and Development, 14, 101-119.
- [Background] McClelland MM, Cameron CE, Connor CM, Farris CL, Jewkes AM, Morrison FJ. Links between behavioral regulation and preschoolers' literacy, vocabulary, and math skills. Dev Psychol. 2007 Jul;43(4):947-59. doi: 10.1037/0012-1649.43.4.947. PMID 17605527
- [Background] Romer D, Betancourt L, Giannetta JM, Brodsky NL, Farah M, Hurt H. Executive cognitive functions and impulsivity as correlates of risk taking and problem behavior in preadolescents. Neuropsychologia. 2009 Nov;47(13):2916-26. doi: 10.1016/j.neuropsychologia.2009.06.019. Epub 2009 Jun 26. PMID 19560477
- [Background] Wilens TE, Martelon M, Fried R, Petty C, Bateman C, Biederman J. Do executive function deficits predict later substance use disorders among adolescents and young adults? J Am Acad Child Adolesc Psychiatry. 2011 Feb;50(2):141-9. doi: 10.1016/j.jaac.2010.11.010. Epub 2011 Jan 6. PMID 21241951
- [Background] Compton, W. M. (2006, June). Enhancing Drug Abuse Prevention Through Type 1 and 2 Translation Research. Paper presented at the Annual Meeting of the Society of Prevention Research, San Antonio, TX.
- [Background] Barth, R. P., & Jonson-Reid, M. (2000). Outcomes after child welfare services: Implications for the design of performance measures. Children and Youth Services Review, 22, 763-787.
- [Background] Courtney ME. The costs of child protection in the context of welfare reform. Future Child. 1998 Spring;8(1):88-103. PMID 9676002
- [Background] Foster, E. M., & Holden, E. W. (2002). Benefit-cost analyses of the child welfare demonstration projects: Understanding the resource implications of the IV-E waivers. Children and Youth Services Review, 24, 431-453.
- [Background] Lee, S., Aos, S., & Miller, M. (2008). Evidence-based programs to prevent children from entering and remaining in the child welfare system: Benefits and costs for washington. Olympia, WA: Washington State Institute for Public Policy.
- [Background] Hoagwood K, Burns BJ, Kiser L, Ringeisen H, Schoenwald SK. Evidence-based practice in child and adolescent mental health services. Psychiatr Serv. 2001 Sep;52(9):1179-89. doi: 10.1176/appi.ps.52.9.1179. PMID 11533391
- [Background] Elliott, D. S. (1998). Blueprints for violence prevention. Boulder, CO: Institute of Behavioral Science, University of Colorado.
- [Background] U.S. Department of Health and Human Services. (2000). Children and mental health. In Mental health: A report of the Surgeon General (DHHS publication No. DSL 2000-0134-P). Washington, DC: U.S. Government Printing Office.
- [Background] U.S. Department of Health and Human Services. (2000). Prevention of violence. In Mental health: A report of the Surgeon General (DHHS publication No. DSL 2000-0134-P). Washington, DC: U.S. Government Printing Office.
- [Background] Chamberlain, P. (1998). Treatment Foster Care. Family Strengthening Series (OJJDP Bulletin NCJ l734211). Washington, DC: U.S. Department of Justice.
- [Background] Reid, J. B., & Eddy, J. M. (1997). The prevention of antisocial behavior: Some considerations in the search for effective interventions. In D. M. Stoff, J. Breiling, J. D. Maser (Eds.), Handbook of antisocial behavior (pp. 343-356). Hoboken, NJ: Wiley.
- [Background] Chamberlain, P., & Reid, J. B. (1987). Parent observation and report of child symptoms. Behavioral Assessment, 9, 97-109.
- [Background] Chamberlain, P., Davis, J. P., Buchanan, R., & Sprengelmeyer, P. (2010). Facilitator Adherence Ratings Unpublished instrument available from Oregon Social Learning Center.
- [Background] Healey, C. V., Bronz, K. D., Fisher, P. A., & Pears, K. C. (2010). KEEP-P Playgroup Implementation Fidelity Checklist. Unpublished instrument available from Oregon Social Learning Center.
- [Background] Gold, M. R., et al. (1996). Identifying and valuing outcomes. In M. R. Gold (Ed.), Cost-effectiveness in health and medicine: Report to U.S. Public Health Service by the Panel on Cost-Effectiveness in Health and Medicine. Washington, DC: U.S. Dept. of Health and Human Services.
- [Background] Brazier J, Czoski-Murray C, Roberts J, Brown M, Symonds T, Kelleher C. Estimation of a preference-based index from a condition-specific measure: the King's Health Questionnaire. Med Decis Making. 2008 Jan-Feb;28(1):113-26. doi: 10.1177/0272989X07301820. Epub 2007 Jul 19. PMID 17641139
- [Background] Dolan P. Developing methods that really do value the 'Q' in the QALY. Health Econ Policy Law. 2008 Jan;3(Pt 1):69-77. doi: 10.1017/S1744133107004355. PMID 18634633
- [Background] Knapp M, Mangalore R. "The trouble with QALYs...". Epidemiol Psichiatr Soc. 2007 Oct-Dec;16(4):289-93. doi: 10.1017/s1121189x00002451. PMID 18333423
- [Background] Lave JR, Frank RG, Schulberg HC, Kamlet MS. Cost-effectiveness of treatments for major depression in primary care practice. Arch Gen Psychiatry. 1998 Jul;55(7):645-51. doi: 10.1001/archpsyc.55.7.645. PMID 9672056
- [Background] Simon GE, Ludman EJ, Rutter CM. Incremental benefit and cost of telephone care management and telephone psychotherapy for depression in primary care. Arch Gen Psychiatry. 2009 Oct;66(10):1081-9. doi: 10.1001/archgenpsychiatry.2009.123. PMID 19805698
- [Background] French MT, Fang H, Fretz R. Economic evaluation of a prerelease substance abuse treatment program for repeat criminal offenders. J Subst Abuse Treat. 2010 Jan;38(1):31-41. doi: 10.1016/j.jsat.2009.06.001. Epub 2009 Jul 23. PMID 19631489
- [Background] Rosenheck R, Kasprow W, Frisman L, Liu-Mares W. Cost-effectiveness of supported housing for homeless persons with mental illness. Arch Gen Psychiatry. 2003 Sep;60(9):940-51. doi: 10.1001/archpsyc.60.9.940. PMID 12963676
- [Background] Farmer, E. M. Z., Angold, A., Burns, B. J., & Costello, E. J. (1994). Reliability of self-reported service use: Test-retest consistency of children's responses to the Child and Adolescent Services Assessment (CASA). Journal of Child and Family Studies, 3, 307-325.
- [Background] Ascher, B. H., Farmer, E. M. Z., Burns, B. J., & Angold, A. (1996). The Child and Adolescent Services Assessment (CASA): Description and psychometrics. Journal of Emotional and Behavioral Disorders, 4, 12-20.
- [Background] Domino ME, Foster EM, Vitiello B, Kratochvil CJ, Burns BJ, Silva SG, Reinecke MA, March JS. Relative cost-effectiveness of treatments for adolescent depression: 36-week results from the TADS randomized trial. J Am Acad Child Adolesc Psychiatry. 2009 Jul;48(7):711-720. doi: 10.1097/CHI.0b013e3181a2b319. PMID 19465880
- [Background] Muthén, L. K., Muthén, B. O. (2010). Mplus user's guide (6th ed.). Los Angeles: CA: Authors.
- [Background] Schafer, J. L. (1997). Analysis of incomplete multivariate data. London, UK: Chapman and Hall.
- [Background] Allison PD. Missing data techniques for structural equation modeling. J Abnorm Psychol. 2003 Nov;112(4):545-57. doi: 10.1037/0021-843X.112.4.545. PMID 14674868
- [Background] Curran PJ, Hussong AM. The use of latent trajectory models in psychopathology research. J Abnorm Psychol. 2003 Nov;112(4):526-44. doi: 10.1037/0021-843X.112.4.526. PMID 14674867
- [Background] Arbuckle, J. L. (1996). Full information estimation in the presence of incomplete data. In G. A. Marcoulides & R. E. Schumacker (Eds.), Advanced structural equation modeling. Mahwah, NJ: Erlbaum.
- [Background] Muthén, L. K., & Muthén, B. O. (2002). How to use a Monte Carlo study to decide on sample size and determine power. Structural Equation Modeling, 9, 599-620.
- [Background] Chamberlain P, Brown CH, Saldana L, Reid J, Wang W, Marsenich L, Sosna T, Padgett C, Bouwman G. Engaging and recruiting counties in an experiment on implementing evidence-based practice in California. Adm Policy Ment Health. 2008 Jul;35(4):250-60. doi: 10.1007/s10488-008-0167-x. Epub 2008 Feb 27. PMID 18302015
- [Background] Drummond, M. F., Sculpher, M. J., Torrance, G. W., O'Brien, B. J., & Stoddart, G. L. (2005). Methods for the economic evaluation of health care programmes. Oxford, UK: Oxford University Press.
- [Background] Foster EM, Connor T. Public costs of better mental health services for children and adolescents. Psychiatr Serv. 2005 Jan;56(1):50-5. doi: 10.1176/appi.ps.56.1.50. PMID 15637192
- [Background] Haddix, A. C., Teutsch, S. M., & Corso, P. S. (Eds.). (2003). A guide to decision analysis and economic evaluation (2nd ed.). New York, NY: Oxford University Press.
- [Background] Edwards RT, Ceilleachair A, Bywater T, Hughes DA, Hutchings J. Parenting programme for parents of children at risk of developing conduct disorder: cost effectiveness analysis. BMJ. 2007 Mar 31;334(7595):682. doi: 10.1136/bmj.39126.699421.55. Epub 2007 Mar 9. PMID 17350965
- [Background] Foster EM, Jones DE. The economic analysis of prevention: an illustration involving children's behavior problems. J Ment Health Policy Econ. 2007 Dec;10(4):165-75. PMID 18166828
- [Background] Hoch JS, Briggs AH, Willan AR. Something old, something new, something borrowed, something blue: a framework for the marriage of health econometrics and cost-effectiveness analysis. Health Econ. 2002 Jul;11(5):415-30. doi: 10.1002/hec.678. PMID 12112491
- [Background] Thompson SG, Barber JA. How should cost data in pragmatic randomised trials be analysed? BMJ. 2000 Apr 29;320(7243):1197-200. doi: 10.1136/bmj.320.7243.1197. No abstract available. PMID 10784550
- [Background] O'Brien BJ, Briggs AH. Analysis of uncertainty in health care cost-effectiveness studies: an introduction to statistical issues and methods. Stat Methods Med Res. 2002 Dec;11(6):455-68. doi: 10.1191/0962280202sm304ra. PMID 12516984
- [Background] O'Brien BJ, Drummond MF, Labelle RJ, Willan A. In search of power and significance: issues in the design and analysis of stochastic cost-effectiveness studies in health care. Med Care. 1994 Feb;32(2):150-63. doi: 10.1097/00005650-199402000-00006. PMID 8302107
- [Background] Knapp M, McCrone P, Fombonne E, Beecham J, Wostear G. The Maudsley long-term follow-up of child and adolescent depression: 3. Impact of comorbid conduct disorder on service use and costs in adulthood. Br J Psychiatry. 2002 Jan;180:19-23. doi: 10.1192/bjp.180.1.19. PMID 11772846
- [Background] Mooney, C. Z., & Duval, R. D. (1993). Bootstrapping: A non-parametric approach to statistical inference. Newbury Park, CA: Sage.
- [Background] Fenwick E, O'Brien BJ, Briggs A. Cost-effectiveness acceptability curves--facts, fallacies and frequently asked questions. Health Econ. 2004 May;13(5):405-15. doi: 10.1002/hec.903. PMID 15127421
- [Background] Little, R. J. A., & Rubin, D. B. (2002). Statistical analysis with missing data (2nd ed.). New York, NY: Wiley.
- [Background] Royston, P. (2004). Multiple imputation of missing values. Stata Journal, 4, 227-241.
- [Background] Royston, P. (2005). Multiple imputation of missing values: Update. Stata Journal, 5, 188-201.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Numbers reported are number of participants (caregivers and their children).
  The "Protocol Enrollment" number (442) differs from the number of participants in the "Started" category (416) due to a control group condition (services as usual) being removed from the study early on. 416 started in the two study conditions (KEEP-P and KEEP-P+)
Groups:
- KEEP-P: The KEEP-P caregiver support groups employ a manualized 12-session, weekly curriculum for foster, kinship, and biological caregivers. Each weekly 2 hour session is structured so that the curriculum content is integrated into group discussions, and primary concepts are illustrated via role-play. Home practice assignments are given weekly and relate to the topics covered during sessions to assist parents in implementing the behavioral procedures taught.
- KEEP-P+: The KEEP-P+ group received the same 12-session, weekly curriculum as the KEEP-P group, and also received an additional video coaching component. The video coaching employs video of caregivers' natural interactions with their child to show ways that they are supporting children's healthy development. It is a simple and practical approach that emphasizes caregivers' strengths and capabilities. It begins with video recordings of a caregiver and child in their home or other natural setting. The film is carefully edited to show brief clips in which the caregiver is engaged in developmentally supportive interactions with the child. At a group coaching session, a coach reviews the edited clips in detail with the caregivers.
Period: Overall Study
Arm/Group | KEEP-P | KEEP-P+
Started | 226 | 190
Completed (Completed post-intervention data collection) | 182 | 164
Not Completed | 44 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KEEP-P | KEEP-P+ | Total
Number analyzed (Participants) | 226 | 190 | 416
Age, Categorical [Count of Participants; unit: Participants] — Population: Numbers are different due to missing data.
  Participants
    number analyzed (Participants) | 216 | 181 | 397
    <=18 years | 107 | 90 | 197
    Between 18 and 65 years | 101 | 90 | 191
    >=65 years | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years]
  Caregivers | 48.62 (11.355) | 45.86 (9.63) | 47.37 (10.669)
  Children | 2.61 (.888) | 2.32 (.633) | 2.48 (.793)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Numbers are different due to missing data.
  Participants
    number analyzed (Participants) | 217 | 181 | 398
    Female | 126 | 114 | 240
    Male | 91 | 67 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 27 | 40
  Not Hispanic or Latino | 169 | 155 | 324
  Unknown or Not Reported | 44 | 8 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 126 | 131 | 257
  More than one race | 40 | 39 | 79
  Unknown or Not Reported | 48 | 16 | 64
Region of Enrollment [Number; unit: participants]
  United States | 226 | 190 | 416

OUTCOME MEASURES:

1. Primary Outcome: Parenting Stress Via Self-report Measure Parenting Stress Index IV (PSI-IV) Short Form
Description: The Parenting Stress Index IV (PSI-IV) Short Form evaluates the magnitude of stress in the parent-child relationship based on the parent's perception of the child's characteristics, the personal characteristics of the parent, and the interaction between the parent and child.
  It is a 5-point Likert scale ranging from "strongly agree" to "strongly disagree" with 36 items. Item 32 is the only item which is reverse coded. For all the other items, higher scores indicate higher levels of stress.
  Total parenting stress score is calculated by summing up scores of all the 36 items, ranging from 36 to 180.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: The number analyzed in the endpoint and change rows is different from the baseline row because we were not able to retain every participant for the post-intervention data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 82 | 84
score on a scale
  Baseline | 80.87 (20.28) | 86.18 (23.83)
  Endpoint: number analyzed (Participants) | 58 | 69
  Endpoint | 74.62 (20.29) | 80.8 (22.76)
  Change: number analyzed (Participants) | 58 | 69
  Change | -5.29 (9.45) | -5.72 (13.97)

2. Primary Outcome: Caregiver's Perceived Sense of Competency in Parenting Via Self-report Measure Parent Sense of Competency Scale (PSOC)
Description: The FOI-adapted Parenting Sense of Competence (PSOC) questionnaire is filled out by the caregiver to assess parents' sense of competence and enjoyment of parenting. This is an adapted version of the PSOC (original PSOC has 17 items, Johnston & Mash, 1989), with 18 items and simplified language for lower reading levels.
  Items are answered on a 4-point Likert scale ranging from "strongly agree" to "strongly disagree." Nine items (#s 2,3,4,5,8,9,13,15 and 17) are reverse coded so that, for all items, higher scores indicate greater parenting self-esteem.
  Total score of parent's perceived sense of competency is calculated by summing up scores of all the 18 items, ranging from 18 to 72.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 81 | 83
score on a scale
  Baseline | 49.42 (5.18) | 49.82 (6.33)
  Endpoint: number analyzed (Participants) | 58 | 68
  Endpoint | 51.6 (5.46) | 50.15 (5.22)
  Change: number analyzed (Participants) | 57 | 67
  Change | 2.14 (3.39) | 0.3 (4.84)

3. Primary Outcome: Observed Level of Developmentally-supportive Parenting Via Observational Measure Parenting Interactions With Children: Checklist of Observations Linked to Outcomes (PICCOLO)
Description: "The Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) is an observational measure which rates developmentally-supportive parenting across four domains: affection, responsiveness, encouragement, and teaching.
  It is a checklist of 29 items reflecting positive parent-child interaction behaviors. Each behavior is rated according to their frequency as 0 (absent, no behavior observed), 1 (barely, minor or emerging behavior) and 2 (clearly, definitive, strong and frequent behavior). Higher scores indicating higher levels of positive parenting.
  PICCOLO total score is calculated by summing up scores of all the 29 items, ranging from 0 to 58. "
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 84 | 86
score on a scale
  Baseline | 42.58 (7.22) | 43.36 (6.65)
  Endpoint: number analyzed (Participants) | 61 | 66
  Endpoint | 42.85 (8.45) | 43.08 (7.65)
  Change: number analyzed (Participants) | 59 | 66
  Change | 0.14 (8.67) | -0.76 (8.57)

4. Primary Outcome: Frequency of Family Routines Via Self-report Measure Family Routines Questionnaire (FRQ)
Description: "The Family Routines Questionnaire (FRQ) is a 28-item measure of the frequency and rated importance of family routines. Scores are calculated based on the how frequent the family's routines are and how important the routines are to them. The frequency of family routines construct was reported in the results.
  To rate each endorsed routine by the frequency of its performance by the family, daily performance is assigned a weight of 3, a somewhat less frequency performance of 3-5 times a week is assigned a weight of 2; and an even less frequent performance of l-2 times a week is assigned a weight of 1. The 'almost never' category is taken to mean that the family does not participate in the particular routine, and it is therefore assigned a value of 0 in computing the total inventory score. By summing up frequency scores of all the 28 items, the total frequency score ranges from 0 to 84. Higher scores indicate higher frequency of family routines."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 83 | 82
score on a scale
  Baseline | 51.66 (11.66) | 50.43 (9)
  Endpoint: number analyzed (Participants) | 60 | 69
  Endpoint | 52.63 (9.79) | 52.09 (9.32)
  Change: number analyzed (Participants) | 59 | 67
  Change | 1.37 (10.34) | 1.3 (6.62)

5. Primary Outcome: Mindful Parenting Via Self-report Measure Interpersonal Mindfulness in Parenting (IEMP)
Description: "The Interpersonal Mindfulness in Parenting (IEMP) scale is a 10-item measure to investigate the quality of interpersonal mindfulness in parenting.
  Items are answered on a 5-point Likert scale ranging from ""never true"" to ""always true"". Four items (#s 1,5,9, and 10) are reverse coded.
  Total score is the sum of all the item scores, ranging from 10 to 50. Higher scores indicate higher quality of Mindful parenting."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 83 | 84
score on a scale
  Baseline | 37.87 (3.33) | 37.17 (4.55)
  Endpoint: number analyzed (Participants) | 59 | 70
  Endpoint | 38.8 (3.36) | 37.56 (4)
  Change: number analyzed (Participants) | 58 | 70
  Change | 0.81 (2.67) | 0.69 (4.03)

6. Primary Outcome: Child Attachment Behaviors Via Caregiver-report Measure Attachment Diary (ADRY)
Description: The Attachment Diary (ADRY) is a 47-item measure in which caregivers report how the child reacts when hurt, frightened, or separated from the caregiver by placing check marks on a behavior list. All the checked behaviors are coded into three categories, proximity seeking/contact maintenance, avoidance, and resistance, to assess individual differences in child's attachment behaviors. Thus, there are no total scores for the ADRY, only subscale scores for the three categories.
  Outcomes include scores for proximity seeking/contact maintenance (range from 0 to 14), scores for avoidance (range from 0 to 18), and scores for resistance (range from 0 to 6), which are generated by counting the number of checked behaviors in corresponding subscales. Higher scores indicate higher levels of behaviors correspondingly.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 83 | 83
score on a scale
  Baseline Proximity | 7.53 (3.89) | 8.42 (3.73)
  Endpoint Proximity: number analyzed (Participants) | 60 | 69
  Endpoint Proximity | 7.75 (3.83) | 7.87 (3.78)
  Change Proximity: number analyzed (Participants) | 59 | 68
  Change Proximity | 0.22 (3.41) | -0.49 (4.17)
  Baseline Avoidance | 1.84 (2.22) | 1.95 (2.19)
  Endpoint Avoidance: number analyzed (Participants) | 60 | 69
  Endpoint Avoidance | 1.78 (2.33) | 2.06 (2.53)
  Change Avoidance: number analyzed (Participants) | 59 | 68
  Change Avoidance | -0.03 (2.15) | -0.04 (2.22)
  Baseline Resistance | 0.72 (1.03) | 0.88 (1.15)
  Endpoint Resistance: number analyzed (Participants) | 60 | 69
  Endpoint Resistance | 0.57 (1.08) | 0.70 (0.99)
  Change Resistance: number analyzed (Participants) | 59 | 68
  Change Resistance | -0.08 (0.95) | -0.21 (1.10)

7. Primary Outcome: Child Internalizing/Externalizing Symptoms and Total Behavior Score Via Caregiver-report Measure Child Behaviour Checklist (CBCL)
Description: The Child Behavior Checklist (CBCL) is a 100-item questionnaire to assess emotional and behavioral problems in children. Caregivers are asked to rate how often their child displayed certain behaviors in the past two months on a 3-point Likert scale (0 = Not True, 1 = Somewhat/Sometimes True, 2 = Very True/Often True).
  Subscales include: Internalizing symptoms - Emotionally Reactive: 21, 46, 82, 83, 92, 97, 99; Anxious/Depressed: 10, 33, 37, 43, 47, 68, 87, 90; Somatic Complaints: 1, 7, 39, 45, 78, 86, 93; Withdrawn: 2, 4, 12, 19, 23, 62, 67, 70, 71, 98 Externalizing symptoms - Attention Problems: 5, 6, 24, 48, 51, 56, 59, 64, 95; Aggressive Behavior: 8, 14, 15, 16, 17, 18, 20, 22, 27, 28, 29, 35, 40, 42, 44, 53, 58, 66, 69, 74, 81, 84, 85, 88, 96 Raw scores for each subscale were calculated by summing up item scores correspondingly and then normalized to T-scores. The means are anchored to 50, with a standard deviation of 10 points. Higher T score indicates more behavior problems.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 85 | 83
T-score
  Baseline | 59.6 (12.13) | 61.65 (11.72)
  Endpoint: number analyzed (Participants) | 62 | 70
  Endpoint | 57.18 (12.44) | 57.47 (12.14)
  Change: number analyzed (Participants) | 62 | 70
  Change | -3.24 (6.95) | -3.76 (6.63)

8. Primary Outcome: Preschool and Kindergarten Behavior Scales (PKBS)
Description: Caregivers perception of their child's behaviors via the Preschool and Kindergarten Behavior Scales (PKBS). Items are on a 4-point scale ranging from "never" to "often." Higher scores indicate more behavior problems.
  PKBS total score (76 items) sum score ranging between 0-228.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total score on scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 80 | 82
total score on scale
  Baseline | 55.86 (19.56) | 54.63 (19.7)
  Endpoint: number analyzed (Participants) | 59 | 69
  Endpoint | 50.6 (21.93) | 52.39 (18.3)
  Change: number analyzed (Participants) | 56 | 67
  Change | -3.44 (10.8) | -3.09 (11.02)

9. Primary Outcome: Parental Stress Via Caregiver-report Measure Parent Daily Report (PDR)
Description: "The Parent Daily Report (PDR) is a caregiver-report measure assessing child behaviour problems and associated parental stress occurring in the past 24 hours. The measure has several versions. The version used in the present research is the Oregon Social Learning Center Community Programs PDR which has 39 questions with only negative child behaviors, targeting to children from 3 to 6 years.
  Caregivers rate each child behavior as 0 = Did Not Occur, 1 = Occurred & Not Stressful, 2 = Occurred & Stressful. The PDR was administered 3 times per wave. For each response, total score of stressful behaviors was calculated by counting the number of behaviors rated as 2 = Occurred & Stressful. Then the three total scores was averaged to get the mean of stressful behaviors (ranges from 0 to 39) as a indicator of parental stress. Higher score indicates higher level of parental stress."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 84 | 84
score on a scale
  Baseline | 6.56 (5.65) | 7.26 (5.36)
  Endpoint: number analyzed (Participants) | 63 | 70
  Endpoint | 4.48 (4.81) | 4.58 (4.11)
  Change: number analyzed (Participants) | 62 | 70
  Change | -1.9 (4.59) | -2.8 (3.98)

10. Primary Outcome: Child Social-emotional Development Via Caregiver-report Measure Ages and Stages Questionnaire: Social-Emotional (ASQ:SE)
Description: "The Ages and Stages Questionnaires: Social-Emotional Development Screening Tool (ASQ:SE) is a caregiver-report questionnaire about children's social-emotional development.
  The ASQ:SE has 29 questions, of which 26 questions are scored from 0-15, the others are open-ended. Therefore the total score (the sum of the 26 item scores) ranges from 0 to 390. Lower scores indicate more pocitive outcomes, i.e. better social-emotional development."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 85 | 86
score on a scale
  Baseline | 121.35 (77.58) | 125.81 (66.21)
  Endpoint: number analyzed (Participants) | 60 | 69
  Endpoint | 105 (74.47) | 119.13 (71.29)
  Change: number analyzed (Participants) | 60 | 69
  Change | -14.33 (33.95) | -2.39 (42.64)

11. Primary Outcome: Observed Level of Child Inhibitory Control Via Delay Choice Paradigm
Description: "In the Delay Choice Paradigm, children were asked to make choices between ""getting one penny/sticker/treat now"" or ""four (or more) to bring home"" for nine times.
  Total score is the total times when the child chooses the ""bring home"" option (ranges from 0 to 9). Higher score indicates better ability for child to delay gratification, i.e. better inhibitory control."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 72 | 75
score on a scale
  Baseline | 4.86 (3.11) | 5.55 (2.91)
  Endpoint: number analyzed (Participants) | 58 | 61
  Endpoint | 5.24 (3.26) | 4.54 (3.5)
  Change: number analyzed (Participants) | 52 | 56
  Change | 0.19 (3.13) | -0.89 (3.41)

12. Primary Outcome: Dimensional Change Card Sort (DCCS)
Description: The total number of phases passed in the DCCS. A phase was passed if 4/6 trials were correct. Children only proceeded to the next phase if they passed the previous phase. 5 phases total. Higher score indicates better executive functioning.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of phases passed
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 78 | 80
number of phases passed
  Baseline | 1.76 (1.43) | 1.61 (1.32)
  Endpoint: number analyzed (Participants) | 60 | 63
  Endpoint | 2.12 (1.54) | 2.05 (1.54)
  Change: number analyzed (Participants) | 58 | 80
  Change | 0.48 (1.29) | 0.43 (1.37)

13. Primary Outcome: Observed Level of Child Inhibitory Control Via Bear/Dragon Task
Description: In the Bear/Dragon Task, children were presented with a "nice bear" and a "mean dragon" and instructed to do what the bear says (e.g., "touch your nose"), but not to do what the dragon says.
  Children's compliance was scored on a 4-point scale on 5 bear trials (0 = failure to move; 1 = a wrong movement; 2 = a partial movement; 3 = a full correct movement) and 5 dragon trials (0 = a full commanded movement; 1 = a partial commanded movement; 2 = a flinch or wrong movement; 3 = no movement). Scores of each trial are summed up to produce a total score ranging from 0 to 30. A higher score indicates better inhibitory control.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 64 | 65
total score
  Baseline | 21.52 (7.58) | 20.42 (8.25)
  Endpoint: number analyzed (Participants) | 50 | 57
  Endpoint | 23.6 (6.81) | 22.42 (7.37)
  Change: number analyzed (Participants) | 43 | 51
  Change | 1.56 (6.41) | 3.24 (8.5)

14. Primary Outcome: Observed Level of Child Working Memory Via Spin the Pots Task
Description: "In the Spin the Pots Task, several visually distinct boxes were arranged on a rotating tray (2.5-year -olds: 8 boxes; 3-year-olds: 9 boxes; 3.5 year olds: 10 boxes; 4-year-olds; 11 boxes). Children watched the experimenter hide colourful stickers inside all but two boxes, cover the boxes with a cloth, and rotate a tray for a few seconds to mark the beginning of a search trial. The cloth was removed and children were instructed to select a box to find a sticker. If a sticker was found, children were allowed to keep it. After each search attempt, the tray was covered and rotated again to mark the beginning of the next search trial. The task was completed once children found all hidden stickers or after the allotted number of trials (2.5-year -olds: 12 trials; 3-year-olds: 14 trials; 3.5 year olds: 16 trials; 4-year-olds; 18 trials).
  Ratio of stickers found to number of trials ranges from 0 to 1. A higher score indicates better working memory."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio of stickers found to trials
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 81 | 79
Ratio of stickers found to trials
  Baseline | 0.58 (.16) | 0.55 (.16)
  Endpoint: number analyzed (Participants) | 60 | 64
  Endpoint | 0.62 (.2) | 0.59 (.18)
  Change: number analyzed (Participants) | 57 | 58
  Change | 0.05 (.22) | 0.06 (.23)

15. Primary Outcome: Silly Animal Categories
Description: Proportion of animals sorted correctly after rule switch. Higher score indicates better executive functioning.
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 76 | 80
proportion correct
  Baseline | 0.64 (.38) | 0.61 (.34)
  Endpoint: number analyzed (Participants) | 56 | 63
  Endpoint | 0.67 (.35) | 0.71 (.31)
  Change: number analyzed (Participants) | 53 | 61
  Change | 0.05 (.33) | 0.1 (0.31)

16. Primary Outcome: Child Executive Function Via Kansas Reflection-Impulsivity Scale for Preschoolers (KRISP)
Description: "The Kansas Reflection-Impulsivity Scale for Preschoolers (KRISP) presents children with a target picture and 4-6 similar pictures. Children were asked to identify an exact match of the target picture.
  Fifteen test trials were administered following a single practice trial. Each item was scored based on the number of incorrect responses, up to 3 errors. Final score is calculated as the number of errors subtracted from the total errors possible (45), ranging from 0 to 45. Higher score indicates better executive functioning."
Time Frame: Change from baseline at endpoint (3-4 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KEEP-P | KEEP-P+
Number analyzed (Participants) | 68 | 67
score on a scale
  Baseline | 35.76 (7.9) | 33.52 (7.78)
  Endpoint: number analyzed (Participants) | 53 | 54
  Endpoint | 37.81 (6.23) | 35.8 (7.6)
  Change: number analyzed (Participants) | 45 | 50
  Change | 2.16 (8.97) | 3.96 (7.55)

ADVERSE EVENTS:
Time Frame: 18 months (or for as long as they were in the study if we lost contact)
Description: This study aims to help caregivers with best practices in parenting, and participants were not exposed to any health risks. Therefore, the potential for participants to be at risk for Serious Adverse Events and All-Cause Mortality is believed to be zero.
Arm/Group | KEEP-P | KEEP-P+
All-Cause Mortality (participants affected / at risk) | 0/226 | 0/190
Serious Adverse Events (participants affected / at risk) | 0/226 | 0/190
Other Adverse Events (participants affected / at risk) | 0/226 | 0/190

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03106636/Prot_SAP_ICF_000.pdf